CLINICAL TRIAL: NCT02413853
Title: PRIMIER*: Randomized Phase II Trial of mFOLFOX6/Bevacizumab With or Without PRI-724 as First Line Treatment for Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy and Bevacizumab With or Without PRI-724 in Treating Patients With Newly Diagnosed Metastatic Colorectal Cancer
Acronym: PRIMIER
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug supply issues
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Prism Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3C-13-3; NCI-2015-00436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 3C-13-3 (Other: USC Norris Comprehensive Cancer Center); R01CA166161 (NIH); P30CA014089 (NIH)
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Adenocarcinoma; Stage IVA Colorectal Cancer; Stage IVB Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — ICG 001; Bevacizumab; Leucovorin; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (PRI-724, mFOLFOX6/bevacizumab) (Experimental): Patients receive CBP/beta-catenin antagonist PRI-724 IV continuously on days 1-7, bevacizumab IV over 30 minutes, leucovorin calcium IV over 2 hours, oxaliplatin IV over 2 hours, and fluorouracil IV over 46 hours on day 8. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: CBP/beta-catenin Antagonist PRI-724; Biological: Bevacizumab; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis
- Arm II (mFOLFOX6/bevacizumab) (Experimental): Patients receive bevacizumab, leucovorin calcium, oxaliplatin, and fluorouracil as in Arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Drug: Fluorouracil; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: CBP/beta-catenin Antagonist PRI-724 — Given IV
  Other Names: PRI-724; Wnt signaling pathway inhibitor PRI-724
  Arms: Arm I (PRI-724, mFOLFOX6/bevacizumab)
Biological: Bevacizumab — Given IV
  Other Names: Avastin; rhuMab-VEGF
Drug: Leucovorin Calcium — Given IV
  Other Names: CF
Drug: Oxaliplatin — Given IV
Drug: Fluorouracil — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well combination chemotherapy and bevacizumab with or without CBP/beta-catenin antagonist PRI-724 (PRI-724) works in treating patients with newly diagnosed colorectal cancer that has spread to other places in the body. Drugs used in chemotherapy, such as leucovorin calcium, oxaliplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as bevacizumab, may block tumor growth in different ways by targeting certain cells. PRI-724 may help stop the growth of cancer cells by blocking the specific signaling pathway that cancer cells need to grow and spread. It is not yet known whether combination chemotherapy and bevacizumab works better with or without PRI-724 in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the progression-free survival in patients with newly diagnosed metastatic colorectal cancer treated with modified fluorouracil, leucovorin calcium, and oxaliplatin 6 (mFOLFOX6)/bevacizumab and PRI-724 vs. mFOLFOX6/bevacizumab alone.

SECONDARY OBJECTIVES:

I. Overall survival, defined as period from time of randomization to death. II. Response rate. III. Determine the incidence and severity of adverse events of PRI-724 administered as a 7-day continuous infusion in patients treated with mFOLFOX6/bevacizumab and PRI-724.

IV. Determine messenger ribonucleic acid (mRNA) expression levels of genes involved in the Wnt pathway (i.e. survivin) by reverse transcriptase-polymerase chain reaction (RT-PCR) in patients treated with mFOLFOX6/bevacizumab and PRI-724 vs. mFOLFOX6/bevacizumab alone both in circulating tumor cells (CTCs) and tumor biopsy specimens.

V. Determine if CTC survivin and stem cell marker expression is consistent and congruent with expression in tumor specimens.

TERTIARY OBJECTIVES:

I. Determine if a correlation exists between Kirsten rat sarcoma viral oncogene homolog (KRAS)/ B-Raf proto-oncogene, serine/threonine kinase (BRAF) mutation status and intratumoral gene expression of the following Wnt related biomarkers: survivin, vascular endothelial growth factor (VEGF), epidermal growth factor (EGF), epidermal growth factor receptor (EGFR), S100 calcium binding protein A4 (S100A4), EPH receptor B2 (EphB2), connexin43, cyclinD1 in patients treated with mFOLFOX6/bevacizumab and PRI-724 vs. mFOLFOX6/bevacizumab alone.

II. Determine the mutational spectrum in colon cancer tissues. III. Determine single nucleotide polymorphism (SNP) profiles in normal and colon cancer tissues.

IV. Determine and describe tumor heterogeneity in colon cancer tissue prior to and during treatment with PRI-724.

V. Determine gene expression signatures, micro RNA (miRNA) signatures, and deoxyribonucleic acid (DNA) methylation signatures as potential predictive and prognostic markers.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive CBP/beta-catenin antagonist PRI-724 intravenously (IV) continuously on days 1-7, bevacizumab IV over 30 minutes, leucovorin calcium IV over 2 hours, oxaliplatin IV over 2 hours, and fluorouracil IV over 46 hours on day 8. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive bevacizumab, leucovorin calcium, oxaliplatin, and fluorouracil as in Arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage IV colorectal adenocarcinoma without any prior systemic treatment
* Signed informed consent prior to initiation of any study-specific procedure or treatment, including consent to provide blood samples for correlative studies and to obtain a tumor biopsy during the study
* Representative tumor tissue specimens (paraffin block preferred)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Able to comply with the protocol, including tissue and blood sampling
* Leukocytes >= 3,000 per mm^3
* Absolute neutrophil count >= 1,500 per mm^3
* Platelet count >= 100,000 per mm^3
* Hemoglobin >= 9 g/dL (may be transfused to maintain or exceed this level)
* Serum creatinine value < upper limit of normal (ULN) or creatinine clearance of >= 60 mL/min according to Cockgroft-Gault formula
* Urine for proteinuria should be < 2 +; patients discovered to have >= 2 + proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours
* Serum total bilirubin < 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 x ULN (< 5 x ULN if there is evidence of hepatic involvement by malignant disease)
* International normalized ratio =< 1.5 and activated prothrombin time =< 1.5 x ULN for patients not receiving anti-coagulation therapy
* The use of full-dose oral or parenteral anticoagulants is permitted as long as the international normalized ratio (INR) or activated partial thromboplastin time (aPTT) is within therapeutic limits (according to the medical standard of the enrolling institution), and the patient has been on a stable dose of anticoagulants for at least two weeks prior to the first study treatment
* Female patients should not be pregnant or breast-feeding
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone hysterectomy or bilateral oophorectomy; OR
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 months)
* Female patients with childbearing potential should agree to use effective, nonhormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgically sterile) during the study and for a period of at least 3 months following the last administration of study drug
* Female patients with an intact uterus (unless amenorrheic for the last 24 months) must have a negative serum pregnancy test within 72 hours prior to administration of any treatment
* Male patients must agree to use effective contraception during the study and for a period of at least 6 months following the last administration of study drugs, even if they have been surgically sterilized
* Patients with treated brain metastases are eligible for study participation; patients may not receive ongoing treatment with steroids at screening; anticonvulsants (at stable dose) are allowed; treatment for brain metastases may be whole-brain radiotherapy, radiosurgery, neurosurgery, or a combination as deemed appropriate by the treating physician; radiotherapy and stereotactic radiosurgery must be completed at least 28 days prior to randomization
* Archival tumor tissue sample (i.e., representative tumor tissue specimen in paraffin block [preferred] or at least 20 unstained slides) must be requested and available prior to study entry
* Patients must have biopsiable tumor and agree to study biopsy

Exclusion Criteria:

* Any prior systemic treatment for metastatic colorectal cancer
* Known hypersensitivity to any of the components of PRI-724, fluorouracil (5-FU), oxaliplatin or bevacizumab
* Adjuvant systemic treatment for colorectal cancer within last 12 months
* Radiotherapy to any site for any reason within 28 days prior to treatment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Sensory peripheral neuropathy > Common Terminology Criteria for Adverse Events (CTCAE) grade 1
* Corrected QT (QTc) interval > 470 msec (females) or > 450 msec (males)
* Active hepatitis B, hepatitis C
* History of arterial thromboembolic events
* History of abdominal fistula formation, gastrointestinal perforation, or abdominal abscess within six months
* History or evidence of inherited bleeding diathesis or coagulopathy with a risk of bleeding
* Patients must not be pregnant or nursing
* Surgery (including open biopsy), significant traumatic injury within 28 days prior to randomization, or anticipation of the need for major surgery during study treatment
* Any hemorrhage or bleeding event >= CTCAE grade 3 within 4 weeks prior to the start of study medication
* Non-healing wound, ulcer, or bone fracture
* Inadequately controlled hypertension (systolic blood pressure [SBP] > 150mmHg, diastolic blood pressure [DBP] > 100mg Hg)
* Renal insufficiency requiring dialysis
* Known positivity for human immunodeficiency virus (HIV)
* Malignancies other than colorectal adenocarcinoma within 5 years prior to treatment, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, and ductal carcinoma in situ treated surgically with curative intent
* Clinically detectable (by physical exam) third-space fluid collections (e.g. ascites or pleural effusion) that cannot be controlled by drainage or other procedures prior to study entry
* Treatment with any other investigational agent, or participation in another investigational drug trial within 28 days prior to randomization
* Minor surgery, including insertion of an indwelling catheter, within 24 hours prior to the first bevacizumab infusion
* Current or recent (within 10 days prior to first dose of bevacizumab) use of aspirin (> 325 mg/day); prophylactic and therapeutic use of anticoagulants is allowed, e.g., warfarin (1 mg once daily [QD]) for catheter prophylaxis and prophylactic low molecular weight heparin (i.e., enoxaparin [40 mg QD])
* Clinically significant (i.e., active) cardiovascular disease (e.g., cerebrovascular accident or myocardial infarction [MI] within 6 months prior to randomization), unstable angina, congestive heart failure (CHF) (New York Heart Association [NYHA] class >= NII), or serious cardiac arrhythmia that is uncontrolled by medication or may interfere with administration of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From time of randomization to time of progression or death on study whichever comes first, assessed up to 2 years
  PFS will be compared between arms by intent-to-treat using Kaplan-Meier curves. The median PFS and 95% confidence interval (CI) will be estimated. Unstratified and stratified hazard ratios and 95% CI will be estimated using the Cox-regression model.

SECONDARY OUTCOMES:
Overall survival (OS) | From time of randomization until death due to any cause, assessed up to 3 years
  OS by arm will be compared using Kaplan-Meier curves and log-rank test.
Overall response rate | Up to 3 years
  Calculated as the ratio of the number of evaluable patients who experienced a confirmed complete response or partial response by Response Evaluation Criteria In Solid Tumors divided by the total number of randomized patients in each arm. 95% Wilson confidence intervals will be constructed. The difference in response rate by arm will be tested using chi-square test or Fisher's exact test whenever appropriate.
Incidence of adverse events evaluated according to the National Cancer Institute CTCAE version 4.0 | Up to 30 days after the last dose of study drugs
Survivin mRNA expression levels | Up to 3 years
  Survivin expression level changes in CTC by cycles will be analyzed by repeated measures analysis of variance.

OTHER OUTCOMES:
KRAS/BRAF mutation status | Baseline
Intratumoral gene expression of Wnt related biomarkers | Up to 3 years
  The change in the gene expression levels prior to and after treatment will be analyzed by the paired t-test, or signed rank test as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Lenz, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States